CLINICAL TRIAL: NCT03426007
Title: Controlled Ovarian Stimulation and Human Uterine Lavage: A Feasibility Study
Brief Title: Controlled Ovarian Stimulation and Human Uterine Lavage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Previvo Genetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TD-2104
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Infertility, Female
Keywords: uterine lavage; intrauterine insemination; embryo; blastocyst; in vivo; superovulation
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Uterine Lavage (Experimental): Embryo recovery from the uterus following either natural cycle (NC)/intrauterine insemination (IUI), or controlled ovarian hyperstimulation (COH)/intrauterine insemination (IUI).
  Interventions: Procedure: Uterine lavage

INTERVENTIONS:
Procedure: Uterine lavage — embryo recovery from the uterus following either natural cycle (NC)/intrauterine insemination (IUI), or controlled ovarian hyperstimulation (COH)/intrauterine insemination (IUI).

SUMMARY:
This is a feasibility study intended to demonstrate the Previvo Uterine Lavage System's ability to recover embryos from the uterus following either natural cycle (NC)/intrauterine insemination (IUI), or controlled ovarian hyperstimulation (COH)/intrauterine insemination (IUI).

DETAILED DESCRIPTION:
The study is a prospective, multi- center, multiple-arm, feasibility study to evaluate the safety and efficacy of the Previvo System in the recovery of embryos.

This study will recruit up to 500 healthy premenopausal volunteers. Subjects will undergo either natural cycle (NC)/intrauterine insemination (IUI), or controlled ovarian hyperstimulation (COH)/intrauterine insemination (IUI) and have the lavage procedure performed 4-6 days post IUI. It is anticipated that embryos recovered will be cryopreserved for future use or donated for future use.

Subjects will be followed up with for up to 30 days after the lavage procedure. All data will be collected on paper CRFs and analyzed by the Principal Investigator and Study Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal female 18-40 years of age
2. Physically healthy and reasonably healthy family medical history
3. Having both ovaries with patent fallopian tubes, no known reproductive problems
4. BMI between 18-35 Kg/m2
5. Presence of a normal uterine cavity as assessed by sonohysterogram (SHG), hysterosalpingogram (HSG), or ultrasound
6. Evidence of normal uterine anatomy that would not prevent the introduction of the lavage catheter.

Exclusion Criteria:

1. History of, or presence of hydrosalpinx
2. Addiction to alcohol and/or narcotics
3. Had radiotherapy or chemotherapy
4. Existence of an ovarian cyst at the beginning of cycle with suspicion of malignancy or a large benign cyst
5. Contraindication for oral contraceptive pills or other study medication
6. Clinically significant abnormal basic metabolic panel lab results
7. Positive test or history of any of the following conditions:

   1. Human immunodeficiency virus (HIV)
   2. Hepatitis B infection
   3. Hepatitis C infection
   4. Syphilis (RPR)
   5. Chlamydial pelvic infection
   6. Gonorrheal pelvic infection.
   7. Positive Pregnancy Test
8. Prior IUD for 60 days or less, or one currently in place
9. Allergic to study materials, supplies and medication
10. Any active, uncontrolled, clinically significant medical condition as determined by the treating principal investigator

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Event Collection | 30-Days
  Assessment of pain during procedure, bleeding experienced during procedure, and infection symptoms experienced subsequent to procedure. Assessment of fluid recovery, fluid loss through cervix, fluid accumulation in the uterus and fluid loss through fallopian tubes.

SECONDARY OUTCOMES:
Recovery of Embryos | 1 Day
  Demonstrate the Previvo Uterine Lavage System's ability to recover embryos from the uterus following either natural cycle (NC)/intrauterine insemination (IUI), or controlled ovarian hyperstimulation (COH)/intrauterine insemination (IUI).

CONTACTS AND LOCATIONS:
Overall Officials: Gheda Sahyun, MA, Study Director — Sponsor GmbH
Locations (1):
- Punta Mita Hospital, Punta de Mita, Nayarit, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Najmabadi S, Rivas JL, Angle MJ, Nadal A, Bastu E, Munne S, Carson SA, Buster JE, Nakajima ST. Human Uterine Lavage: First Live Births from In Vivo Conceived Genetically Screened Blastocysts. Adv Ther. 2023 May;40(5):2534-2541. doi: 10.1007/s12325-023-02486-1. Epub 2023 Mar 29. PMID 36988819
- [Derived] Munne S, Nakajima ST, Najmabadi S, Sauer MV, Angle MJ, Rivas JL, Mendieta LV, Macaso TM, Sawarkar S, Nadal A, Choudhary K, Nezhat C, Carson SA, Buster JE. First PGT-A using human in vivo blastocysts recovered by uterine lavage: comparison with matched IVF embryo controlsdagger. Hum Reprod. 2020 Jan 1;35(1):70-80. doi: 10.1093/humrep/dez242. PMID 31886877